CLINICAL TRIAL: NCT01169467
Title: Cerebral Perfusion Pressure Using Precedex and Other Sedatives
Acronym: C3PO
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: Hospira, now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Pro00018317
Record Dates: First submitted 2010-07-22; First posted 2010-07-26 (Estimated); Results first posted 2015-11-02 (Estimated); Last update posted 2015-11-02 (Estimated); Status verified 2015-10

CONDITIONS: Endotracheal Intubation; Continuous IV Sedation; ICP Monitoring
MeSH Terms: interventions — Standard of Care; Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard-of-Care plus Precedex (Active Comparator): Subjects who are treated with dexmedetomidine (Precedex) in addition to the standard of care sedation regiment.
  Interventions: Drug: Standard-of-Care plus Dexmedetomidine
- Standard-of-Care (Placebo Comparator): Subjects who are treated with the standard of care sedation regiment only.
  Interventions: Other: Standard-of-Care

INTERVENTIONS:
Drug: Standard-of-Care plus Dexmedetomidine — Subjects who are treated with dexmedetomidine (Precedex) in addition to the standard of care sedation regiment
  Other Names: Precedex
  Arms: Standard-of-Care plus Precedex
Other: Standard-of-Care — Subjects who are treated with the standard of care sedation regiment only.
  Arms: Standard-of-Care

SUMMARY:
The purpose of this study is to examine the effects of using dexmedetomidine (Precedex) in addition to the current standard-of-care for sedation.

DETAILED DESCRIPTION:
Primarily, this study seeks to explore whether there is a difference in mean arterial pressure (MAP) variability, incidence of intracranial hypertension, intracranial pressure (ICP) variability, cerebral perfusion pressure (CPP) and Cerebrovascular pressure reactivity index (PRx) in two groups of subjects.

Patients must be submitted to the ICU and be endotracheally intubated and receiving mechanical ventilation with continuous IV sedation for less than 24 hours after recruitment into the study.

ELIGIBILITY:
Inclusion Criteria:

* Admitted to Duke University Neuro Critical Care Unit (NCCU)
* Adult (18 years of age or older)
* Expected Mechanical Ventilation for >48 hours with sedation
* Intraventricular catheter in situ

Exclusion Criteria:

* Hypersensitivity to study drugs
* Prisoners
* Moribund state or death expected within 24 hours
* Surgery planned within 24 hours of subject enrollment
* Receiving study drug, Precedex, prior to entering study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2009-10; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Keith Dombrowski, MD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

REFERENCES:
- [Background] Lazaridis C, DeSantis SM, Smielewski P, Menon DK, Hutchinson P, Pickard JD, Czosnyka M. Patient-specific thresholds of intracranial pressure in severe traumatic brain injury. J Neurosurg. 2014 Apr;120(4):893-900. doi: 10.3171/2014.1.JNS131292. Epub 2014 Feb 7. PMID 24506248

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 89 subject signed consent, 5 subjects screen failed.
Period: Overall Study
Arm/Group | Standard-of-Care Plus Precedex | Standard-of-Care
Started | 44 | 40
Completed | 37 | 36
Not Completed | 7 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard-of-Care Plus Precedex | Standard-of-Care | Total
Number analyzed (Participants) | 44 | 40 | 84
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 38 | 32 | 70
  >=65 years | 6 | 8 | 14
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 13 | 30
  Male | 27 | 27 | 54
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 1 | 3
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 10 | 15 | 25
  White | 32 | 24 | 56
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 2 | 4
  Not Hispanic or Latino | 42 | 38 | 80
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Variability of Intracranial Pressure (ICP)
Description: Variability of intracranial pressure was assessed and listed as the standard deviation of all measurements within 24 hours. Variability was assessed and listed as the standard deviation of all measurements within 24 hours
Time Frame: Baseline to 24 hours
Population: Everyone who completed the trial was included except for fourteen subjects had incomplete data and could not be included in this analysis.
Measure: Mean (Standard Error); unit: mmHg
Arm/Group | Standard-of-Care Plus Precedex | Standard-of-Care
Number analyzed (Participants) | 34 | 25
mmHg | 5.66 (0.63) | 5.61 (0.64)

2. Primary Outcome: Change in Pressure Reactivity Index (PRx)
Description: Using computational methods, the PRx was determined by calculating the correlation coefficient between 20 consecutive, time-averaged data points (60-second periods) of ICP and Arterial Blood Pressure (ABP).
  A positive PRx correlation suggests impaired cerebrovascular pressure reactivity, that is, passive transmission of changes in ABP to ICP. A negative PRx correlation indicates good pressure reactivity. Any change in ABP produces inverse changes in ICP.
Time Frame: Baseline to 24 hours
Population: Everyone who completed the trial was included except for nineteen subjects had incomplete data and could not be included in this analysis.
Measure: Mean (Standard Error); unit: Pressure Reactivity Index
Arm/Group | Standard-of-Care Plus Precedex | Standard-of-Care
Number analyzed (Participants) | 32 | 22
Pressure Reactivity Index | .64 (.02) | .66 (.02)
Statistical Analysis 1: Comparison: Standard-of-Care Plus Precedex vs Standard-of-Care; Test type: Superiority or Other; p = 0.395, t-test, 2 sided

3. Secondary Outcome: Amount of Sedative/Analgesic Used During Treatment in Patients With Secondary Brain Injury
Description: Improved physiologic Response. A lower use of sedatives or analgesic during treatment would be considered an improved physiologic response. An increase in the use of sedatives or analgesic during treatment would be considered a worse physiologic response.
Time Frame: 24 hours
Population: Everyone who started the trial was included except for one subject had incomplete data and could not be included in this analysis.
Measure: Mean (Standard Error); unit: mg/ml
Arm/Group | Standard-of-Care Plus Precedex | Standard-of-Care
Number analyzed (Participants) | 44 | 39
mg/ml | 155.4 (23.3) | 213.1 (26.3)

4. Secondary Outcome: Cerebral Perfusion Pressure Changes in Patients With Secondary Brain Injury
Description: Improved physiologic Response. A higher cerebral perfusion pressure during treatment would be considered an improved physiologic response. A lower cerebral perfusion pressure during treatment would be considered a worse physiologic response.
Time Frame: Baseline to 24 hours
Population: as for outcome 1
Measure: Mean (Standard Error); unit: mmHg
Arm/Group | Standard-of-Care Plus Precedex | Standard-of-Care
Number analyzed (Participants) | 34 | 25
mmHg | 11.5 (.63) | 12.3 (.74)

5. Secondary Outcome: Mean Arterial Blood Pressure (MAP) Variability in Patients With Secondary Brain Injury
Description: Improved physiologic Response. A lower variability of mean Arterial Blood pressure during treatment would be considered an improved physiologic response. A higher variability of mean Arterial Blood pressure during treatment would be considered a worse physiologic response. Variability was assessed and listed as the standard deviation of all measurements within 24 hours.
Time Frame: Baseline to 24 hours
Population: Everyone who started the trial was included except for seventeen subjects had incomplete data and could not be included in this analysis.
Measure: Mean (Standard Error); unit: mmHg
Arm/Group | Standard-of-Care Plus Precedex | Standard-of-Care
Number analyzed (Participants) | 39 | 28
mmHg | 12.30 (0.73) | 13.8 (1.44)

ADVERSE EVENTS:
Arm/Group | Standard-of-Care Plus Precedex | Standard-of-Care
Serious Adverse Events (participants affected / at risk) | 1/44 | 0/40
Other Adverse Events (participants affected / at risk) | 0/44 | 0/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard-of-Care Plus Precedex (N=44) | Standard-of-Care (N=40)
Death (Withdrawal of Life Support) (General disorders) | 1 (1) | 0 (0) — Family decided to withdraw support on the patient during study period.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No